CLINICAL TRIAL: NCT05318495
Title: A Dual Tandem Study Comparing the Adenoma Detection and Miss-rate of SC to That of Artificial Intelligence (CAD-EYE) Aided Colonoscopy and to That of Artificial Intelligence (CAD-EYE) and G-EYE® Aided Colonoscopy.
Brief Title: A Dual Tandem Study - SC vs. CAD-EYE vs. CAD-EYE With G-EYE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Horst Schmidt Klinik GmbH (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Ralf Kiesslich, Prof., Dr. Horst Schmidt Klinik GmbH
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Dual Tandem
Record Dates: First submitted 2022-03-29; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Adenoma; Colo-rectal Cancer
MeSH Terms: conditions — Adenoma; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Colonoscopy+CAD-EYE followed by Standard Colonoscopy (Experimental): CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
  The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE
- Standard Colonoscopy followed by Standard Colonoscopy+CAD-EYE (Active Comparator): CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
  The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE
- Standard Colonoscopy+CAD-EYE+G-EYE followed by Standard Colonoscopy (Experimental): CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
  The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
  The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning.
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE; Device: G-EYE
- Standard Colonoscopy followed by Standard Colonoscopy+CAD-EYE+G-EYE (Active Comparator): CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
  The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
  The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning.
  Interventions: Device: Standard Colonoscopy; Device: CAD-EYE; Device: G-EYE

INTERVENTIONS:
Device: Standard Colonoscopy — The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
Device: CAD-EYE — CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
Device: G-EYE — The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning.
  Arms: Standard Colonoscopy followed by Standard Colonoscopy+CAD-EYE+G-EYE; Standard Colonoscopy+CAD-EYE+G-EYE followed by Standard Colonoscopy

SUMMARY:
Single-center, four-arm dual-tandem, randomized, open-label study involving the following devices:

1. The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
2. CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
3. The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning.

DETAILED DESCRIPTION:
Single-center, four-arm dual-tandem, randomized, open-label study involving the following devices:

1. The Standard Colonoscope is a high-definition colonoscope employing advanced optical filtering and enhancement techniques - blue light imaging (BLI) and linked color imaging (LCI).
2. CAD-EYE is an artificial intelligence software, used in real-time during the colonoscopy procedure for aiding the identification and characterization of polyps and adenomas.
3. The G-EYE® balloon is a reusable (reprocessable) balloon permanently installed on the distal tip of a standard colonoscope, and is also intended to assist in flattening colonic folds and control the colonoscope's field of view and tip positioning.

Total of up to 372 patients will be randomized,186 to each of the two tandems

ELIGIBILITY:
Inclusion Criteria:

1. Screening and surveillance population for Adenoma and CRC.
2. The patient must understand and sign a written informed consent for the procedure.

Exclusion Criteria:

1. Subjects with inflammatory bowel disease;
2. Subjects with a personal history of hereditary polyposis syndrome;
3. Subjects with suspected chronic stricture potentially precluding complete colonoscopy;
4. Subjects with diverticulitis or toxic megacolon;
5. Subjects with prior colonic surgery (exclusion appendectomy)
6. Subjects with a history of radiation therapy to abdomen or pelvis;
7. Pregnant or lactating female subjects;
8. Subjects who are currently enrolled in another clinical investigation.
9. Subjects with current oral or parenteral use of anticoagulants, not considered eligible by the investigator.
10. Subjects with recent (within the last 3 mounts) coronary ischemia or CVA (stroke)
11. Any patient condition deemed too risky for the study by the investigator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Additional adenoma detection yield | 6 weeks
  additional adenoma detection yield (represented by the miss rate) of CAD-EYE and G-EYE® colonoscopy over standard coloscopy compared to the additional adenoma detection yield of CAD-EYE aided colonoscopy over standard colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Kiesslich, Prof., Principal Investigator — Helios Dr. Horst Schmidt Kliniken Wiesbaden
Locations (1):
- Helios Dr. Horst Schmidt Kliniken, Wiesbaden, Germany